CLINICAL TRIAL: NCT01148485
Title: Community-acquired Methicillin-Resistant Staphylococcus Aureus Carriage Among Athletes: a Study in Limousin. : CA-MRSA
Brief Title: Community-acquired Methicillin-Resistant Staphylococcus Aureus Carriage Among Athletes
Acronym: PSARM-S
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I09016
Record Dates: First submitted 2010-06-16; First posted 2010-06-22 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2010-06

CONDITIONS: Staphylococcus Aureus
Keywords: - Staphylococcus aureus Carriage among Athletes
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Nasal, throat, inguinal and skin lesions swab samples will be performed — Nasal, throat, inguinal and skin lesions swab samples will be performed

SUMMARY:
There are only very few data about the prevalence of CA-MRSA in France and no in athletes. In USA, the clone USA300 is widely disseminated and in Europe the clone ST80 predominates. The aim of the study was to study the carriage of S. aureus in athletes in a French county (Limousin) and to evaluate the proportion of CA-MRSA. The athletes will be met during their training, each one will fill-in a clinical information questionnaire. Nasal, throat, inguinal and skin lesions swab samples will be performed. The antibiotic susceptibility profile of the Staphyloccocus aureus strains isolated will be performed as well as the detection of the PVL gene. Strains will also be typed by different molecular methods (PGFE (Pulsed Gel Field Electrophoresis), SCCmec type (Staphylococcal Chromosome Cassette mec), and MLST (MultiLocus Sequence Typing)). The CIC (Clinical Investigation Center) of the Limoges University Hospital will be in charge of the inclusions of the athletes. The sample analysis will be centralized and performed at the Laboratory of Bacteriology of the Limoges University Hospital. A Clinical Research Officer of the Limoges University Hospital will be in charge of the survey of the study and will organize monthly meetings with all the participants of the study.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (over 18),
* belonging to a sport club of Limousin, practicing rugby, wrestling, basket-ball, volley-ball, hand-ball, fence, martial art, football, weight lifting, and base-ball.
* Patient having signed in a free way and lit his consent to participate in this study

Exclusion Criteria:

* clinical information questionnaire not possible to fill,
* swab sample not possible to realize.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Athletes of Limousin practicing sport.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Presence of Methicillin-Resistant Staphylococcus aureus in the samples. | 1 year
  An athlete is defined as a carrier if at least one strain of Staphylococcus aureus is isolated from one of these samples.
  A MRSA carrier is defined if the resistance to methicillin has been found for the S. aureus strain isolated in the patient.

SECONDARY OUTCOMES:
Comparison of the MRSA prevalence in athletes according to the sport | 1 year
  Comparison of the MRSA prevalence in athletes according to the sport.A strain is considered as PVL positive if the gene encoding the PVL was detected by PCR.

REFERENCES:
- [Derived] Couve-Deacon E, Postil D, Barraud O, Duchiron C, Chainier D, Labrunie A, Pestourie N, Preux PM, Francois B, Ploy MC. Staphylococcus Aureus Carriage in French Athletes at Risk of CA-MRSA Infection: a Prospective, Cross-sectional Study. Sports Med Open. 2017 Aug 16;3(1):28. doi: 10.1186/s40798-017-0094-z. PMID 28815486